CLINICAL TRIAL: NCT04514133
Title: The I-ACTED Study: Testing the Causal Effects of a Civic Engagement Intervention on Health and Wellbeing Among Youth
Brief Title: Testing the Causal Effects of a Civic Engagement Intervention on Health and Wellbeing Among Youth (I-ACTED)
Acronym: I-ACTED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00066103
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Wellness 1; Social Interaction; Health Attitude
Keywords: civic engagement; health; social wellbeing; behavioral health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Action Civics program (Experimental): Students in this arm will take part in an Action Civics (AC) program. AC delivers action civics programming to young people from diverse backgrounds nationwide. AC offers a school-based action civics curriculum in which classes collectively choose a local issue, learn strategies and skills for taking civic action, develop an action plan, and take action on their selected local issue. Students, as a class, tackle topics ranging from health-related (e.g., health of school lunches) to safety-related (e.g. lack of crosswalks) to community social issues (e.g., community-police relations).
  Interventions: Behavioral: Participating in Action Civics program
- No Action Civics program (No Intervention): Students in this arm will receive no intervention.

INTERVENTIONS:
Behavioral: Participating in Action Civics program — Students in school classrooms participating in Action Civics program
  Arms: Action Civics program

SUMMARY:
The purpose of this research is to understand how participating or not participating in an action civics curriculum may affect the health and wellbeing of young people. Participants will be chosen from students who attend certain schools that choose to participate in the action civics curriculum. Participation in this research involves completing surveys during class time in the Spring and Fall 2021-2022 semesters and then completing online surveys outside of class in the future.

DETAILED DESCRIPTION:
Equal access to civic resources, such as opportunities for civic engagement and connections to one's community, are an important part of a culture of health. Meaningful experiences in civic engagement and community connectedness are transformative for young people - especially for youth from marginalized backgrounds, who often feel voiceless and excluded from decision-making in civic and social institutions. Theories and correlational evidence point to positive associations between civic engagement (e.g., volunteering, voting, and feelings of civic empowerment) and better mental, physical, and behavioral health and wellbeing. Meaningful civic engagement experiences may have an especially powerful effect on health and wellbeing for those from traditionally marginalized backgrounds. However, causal pathways between civic interventions, civic outcomes, and health and wellbeing outcomes among are not firmly established. Further, how civic engagement and sense of community affect health and wellbeing outcomes are unknown, and questions remain about for whom these effects may be especially beneficial. In this study, we ask whether an established civic intervention called Action Civics affects civic engagement and sense of community, and subsequently affects health and wellbeing among youth. To build on these observational findings, the study team will: (a) examine the causal links between youth civic engagement and sense of community and health, and (b) test whether an established school-based, civic engagement intervention can affect individual health and wellbeing and equity outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled Middle or High School student
* Enrolled in a course with a teacher from a school participating in the study

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1659 (Actual)
Dates: Start 2021-06-24 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Youth Inventory of Involvement (activism, political engagement, and leadership items) | Baseline
  Questionnaire measures civic engagement using a Likert scale (1-5) with higher composite scores indicating more involvement in each domain
Youth Inventory of Involvement (activism, political engagement, and leadership items) | 4-6 month following baseline
  Questionnaire measures civic engagement using a Likert scale (1-5) with higher composite scores indicating more involvement in each domain
Youth Inventory of Involvement (activism, political engagement, and leadership items) | 1 year following baseline
  Questionnaire measures civic engagement using a Likert scale (1-5) with higher composite scores indicating more involvement in each domain

SECONDARY OUTCOMES:
Community Connection Scale | baseline, 4-6 month following baseline, 1 year following baseline
  Questionnaire measures sense of community using a Likert scale (1-5) with higher scores indicating higher sense of community. Based on from the California Healthy Kids Survey.
Questionnaire from the National Longitudinal Study of Adolescent to Adult Health | baseline, 4-6 month following baseline, 1 year following baseline
  Questionnaire measures physical and mental health and wellbeing. Response options vary from 4-6 levels for the scales; higher numbers indicate better health.

OTHER OUTCOMES:
Center for Epidemiological Studies Depression (CES-D) | baseline, 4-6 month following baseline, 1 year following baseline
  CES-D measures depressive symptoms using a 1-4 range (1=Rarely or none of the time, 2=Some or a little of the time, 3=Occasionally or a moderate amount of time, 4=All of the time). Higher scores CES-D suggest a greater presence of depressive symptoms.
Tobacco, Alcohol, Prescription medication, and other Substance use Tool part 2 (TAPS- 2) | baseline, 4-6 month following baseline, 1 year following baseline
  Behavioral health symptoms will be measured using adapted items from part 2 of the TAPS questionnaire using a 1-4 range (1=never, 2=once or twice, 3=monthly, 4=weekly or more). Scores on these questions generate a risk level per substance endorsed, based on a range of possible scores per substance.
The World Health Organization- Five Well-Being Index (WHO-5) | baseline, 4-6 month following baseline, 1 year following baseline
  WHO5 measures general wellbeing. Responses ranges from 0-25, with 25 representing best possible quality of life.
Social wellbeing-School Absences | baseline, 4-6 month following baseline, 1 year following baseline
  Responses are counted as a continuous variable (number of class days missed) to generate a value.
Social wellbeing-Purpose tool | baseline, 4-6 month following baseline, 1 year following baseline
  Items measure future aspirations/goals using a Likert scale (1-5) with higher composite scores indicating better social wellbeing.

CONTACTS AND LOCATIONS:
Overall Officials: Parissa J Ballard, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballard PJ, Cohen AK, Littenberg-Tobias J. Action Civics for Promoting Civic Development: Main Effects of Program Participation and Differences by Project Characteristics. Am J Community Psychol. 2016 Dec;58(3-4):377-390. doi: 10.1002/ajcp.12103. PMID 27982470
- [Background] Ballard PJ, Hoyt LT, Pachucki MC. Impacts of Adolescent and Young Adult Civic Engagement on Health and Socioeconomic Status in Adulthood. Child Dev. 2019 Jul;90(4):1138-1154. doi: 10.1111/cdev.12998. Epub 2018 Jan 23. PMID 29359473
- [Derived] Cohen AK, Fitzgerald JC, Trejo G, Yalif IU, Wesson PD, Wolfson M, Ballard PJ. The I-ACTED study (investigating action civics training through an experimental design): a cluster randomized controlled trial of a school-based action civics education intervention on adolescent wellbeing. BMC Public Health. 2025 Oct 16;25(1):3513. doi: 10.1186/s12889-025-24838-y. PMID 41102741